CLINICAL TRIAL: NCT04576403
Title: Heated Mittens for Patients With Hand Osteoarthritis: a Randomized Controlled Trial
Brief Title: Heated Mittens for Patients With Hand Osteoarthritis
Acronym: HOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cecilie Bartholdy (Other)
Responsible Party: Sponsor-Investigator, Cecilie Bartholdy, Investigator, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 143 HOT
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hand Osteoarthritis
Keywords: mittens; heat; hand osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to either intervention og control group by use of a randomization list
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A designated person will number the all mittens using a randomization list. The rest of the study personnel (care provider, investigator, outcome assessor) will thereby not be aware of which mittens that functions and which that do not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Activated mittens
  Interventions: Device: activated mittens
- Control group (Sham Comparator): Deactivated mittens
  Interventions: Device: deactivated mittens

INTERVENTIONS:
Device: activated mittens — activated mittens (with electronic heat)
  Arms: Intervention group
Device: deactivated mittens — deactivated mittens (without electronic heat)
  Arms: Control group

SUMMARY:
The primary objective of this trial is to assess the efficacy of an intervention with heated mittens in patients with hand osteoarthritis (HOA).

The joints of the hands are some of the most commonly joints affected by osteoarthritis, together with hip and knee joints. The prevalence increases with age and as the elderly population is growing so will the number of persons with HOA.

The primary symptoms for HOA are reduced function, stiffness and pain, with function being the most limiting factor for the patients.

Pharmacological treatments have some effect. Non-pharmacological treatments (such as exercise) have been investigated in a limited number of studies with overall minimal effect on the primary symptoms. In the earlier days the use of heating interventions, such as paraffin bath, was common treatment for patients with arthritis. During the last decades a shift from heating to exercise oriented treatment has occurred, however seemingly with limited effect on the primary symptoms. American College of Rheumatology (ACR) newest published guideline for the management of HOA (2020) recommend heating as a treatment among others but without scientific sound evidence for effect.

The hypothesis is that heated mittens worn at least 15 minutes every day for six weeks has a beneficial effect on physical function in patient with HOA when compared to placebo mittens (heat deactivated).

This study is designed as a randomized controlled trial with two parallel groups (1:1) and physical function of the hand as primary endpoint after six weeks.

The plan is to include 200 patients with HOA for this study. The intervention group will receive mittens with functioning heating elements; the control group will receive mittens without a functioning heating element. All participants are asked to wear the mittens for 6 weeks, 15 minutes each day.

The primary endpoint is change in physical function of the hand, measured with the Australian/Canadian Osteoarthritis Hand Index (AUSCAN).

DETAILED DESCRIPTION:
The primary objective of this trial is to assess the efficacy of an intervention with heated mittens in patients with hand osteoarthritis (HOA).

The joints of the hands are some of the most commonly joints affected by osteoarthritis, together with hip and knee joints. Approximately 40% of adults have both self-reported and X-ray conformed signs of HOA. The prevalence increases with age and as the elderly population is growing so will the number of persons with HOA.

HOA is a heterogeneous disease with varying levels of symptoms and joint involvement. The most frequently affected joints are the carpometacarpal (CMC) 1 joints together with the distal interphalangeal (DIP), less frequent the proximal interphalangeal (PIP) joints. The primary symptoms are reduced function, stiffness and pain.

Pharmacological treatments have limited effect. Non-pharmacological treatments (such as exercise) have been investigated in a limited number of studies with overall minimal effect on the primary symptoms. In the earlier days the use of heating interventions, such as paraffin bath, were common treatment for patients with arthritis. During the last decades a shift from heating to exercise oriented treatment have occurred, however seemingly with limited effect on the primary symptoms. American College of Rheumatology (ACR) newest published guideline for the management of HOA (2020) recommend heating as a treatment among others but without scientific sound evidence for effect.

An interview have been conducted at the Parker Institute with people suffering from HOA and all agreed that head was their preferred treatment for symptom reduction. They also stated that heat could reduce stiffness of the fingers. Heating therapy is assumed to provide analgesic effect and decrease muscle tonicity. Two studies have investigated the sort term effect of heat wrap therapy on low back and wrist pain compared to ibuprofen or placebo medication, respectively. In both studies the effect of the heat wrapping therapy was superior to the control group in reducing pain and increasing motion. This suggests that there is a short-term effect of heating therapy in musculoskeletal conditions.

The inflammation level in HOA fluctuates it therefore could be argued that heating therapy may reinforce present inflammation and should be avoided during flares. However, in persons with rheumatoid arthritis heat do not seem to increase the inflammation markers in the synovial tissue.

Studies assessing the potential benefits of non-pharmacological treatments of HOA are scares and both ACR (American College of Rheumatology), EULAR (European League against Rheumatism) and OARSI (Osteoarthritis Research Society International) recommend exploration of this area.

Thus, it is relevant to develop and implement treatment strategies for the management of HOA in order to optimize current treatment strategies.

Based on previous treatment strategies and recent recommendations it seems relevant to investigate if a daily intervention with warm mittens can help reduce pain, improve function and reduce stiffness in patients with HOA.

The aim of this randomized controlled study is to assess the effect of heated mittens after 6 weeks on physical function in patients with HOA.

Heated mittens worn at least 15 minutes every day for six weeks has a beneficial effect on physical function in patient with HOA when compared to placebo mittens (heat deactivated).

STUDY DESIGN This study is designed as a randomised controlled trial with two parallel groups and physical function of the hand as primary endpoint after six weeks.

For each study participant, participation is 6 weeks with clinical assessments at baseline and after 6 weeks.

The number of study participants to be randomised for this study is 200 based on a sample size calculation (see section 14.1). Randomised participants who withdraw during study participation or who are prematurely terminated will not be replaced.

Randomization lists will be computer-generated based upon permuted random blocks of variable size (2 to 6 in each block). The allocation ratio will be 1:1 stratified for the following baseline conditions:

A. CMC 1 OA B. Grip strength

The investigators, outcome assessors, and participants will be blinded to treatment allocation.

The persons performing the phone calls at week 2 and 4 will not be blinded to the allocation.

The HOT intervention consists of a pair of mittens with heating elements. The mittens are produced by Nordic Heat Aps, Denmark. The intensity of the heat can be adjusted by use of a button placed at the dorsal side of the mittens. The mittens have three intensities: red=max, yellow=medium and green=minimum.

The participants are instructed to wear the mittens at least 15 minutes every day, preferably in the morning, for six weeks. If the participants want to use the mittens several times per day or longer than 15 minutes they can. Participants will be instructed to fill out a diary during the intervention period containing the following information; number of times per day they wear the mittens, duration of each wear-time, and intensity level.

Two batteries are placed in the bottom of the mittens with a wire connecting them to the heating element. The batteries must be charged every day, using a charger. In addition to the mittens all participants will receive three pairs of thin cotton gloves (Abena A/S, Aabenraa, Denmark) to use under the mittens for better distribution of the heat.

The mittens, charger, cotton gloves, and diary will be handed out at the baseline visit, after randomization, together with oral and written instructions.

Participants in the control group will receive the same type of mittens but with the heating element being deactivated. Further they will receive cotton gloves to wear underneath the mittens. Both groups will receive the same oral and written instructions on who to use the mittens and all will be instructed to fill out a diary. Participants in both groups will receive a phone call at week 2 and 4 to maintain compliance.

Statistics Sample size A sample size of 200 in total will provide strong statistical power to detect differences between groups in favour of heated mittens. For a two-sample pooled t-test of a normal mean difference with a two-sided significance level of 0.05 (P<0.05), assuming a common standard deviation of 19 AUSCAN-function points (0-100 scale), a total sample size of 180 assuming a balanced design has a power of 80.2% to detect a mean difference of 8 AUSCAN-function points (corresponding to a small effect size of 0.42). To account for dropouts, 200 patients will be included.

Primary analysis population The intention to treat (ITT) population consist of all randomized patients irrespective of whether the patient actually received study intervention or the patient's compliance with the study protocol, in the treatment group to which the participant was assigned at randomisation. A patient will be considered randomised as soon as a treatment is assigned.

Statistical approach A statistical analysis plan that describes the details of the planned statistical analyses will be produced before last patient's last visit.

Assessments of changes from baseline and construction of confidence intervals (CI) for continuous measures will be based on a repeated measures analysis of covariance (ANCOVA; including group as the main factor and baseline measure as covariate). Superiority will be claimed if the computed 95% CI of the estimated group difference in the change from baseline in the AUSCAN does not include 0 in the ITT population. All statistical tests will be two-sided and statistical significance will be claimed if the computed p-value is equal to or less than 0.05.

Case report forms (CRF) The study will use electronic case report forms (eCRF) using an in-house database created specifically to this trial by the Parker Institutes database manager. To additional program will be used to capture the questionnaire registrations electronically: RedCap will be used to supply data from home (AUSCAN send at week 2 and 4), Cirkeline will be used to supply data from the study visits (baseline, week 6).

In addition to the eCRF a paper based CRF is created to allow for on-the-go registration of participants at the clinic. An investigator will be responsible for the transfer of data from the CRF to eCRF during the trial period.

At the end of the trial, all data will be merged and stored in the in-house database. The in-house database meets all regulatory standards and allows management of all activities related to clinical trials that ensures optimal resource use and safety according to good clinical practice and data protection legislation.

Quality assurance All data will be entered into a study database for analysis and reporting. Any data captured electronically will be stored electronically in a separate database according to standard procedures at The Parker Institute. Upon completion of data entry, the databases will be checked to ensure acceptable accuracy and completeness. System backups and record retention for the study data will be consistent with The Parker Institute standard procedures.

Data protection and regulation The study will be conducted in accordance with the Data Protection Act and follow the General Data Protection Regulation. The study data management and data security procedures are approved by the Regional Knowledge Centre on Data Protection Compliance (videnscenter for dataanmeldelser i Region Hovedstaden) on behalf of the Danish Data Protection agency.

ELIGIBILITY:
Inclusion Criteria:

1. HOA with fulfillment of the ACR criteria:

   a. Hand pain, aching or stiffness on most days the previous 4 weeks

   And at least 3 of the following features:
   * Hard tissue enlargement of ≥2 of the 10 selected joints*
   * Hard tissue enlargement of ≥2 of the 10 DIP joints
   * Fewer than 3 swollen metacarpophalangeal (MCP) joints
   * Deformity of at least 1 of 10 selected joints* *The 10 selected joints are the second and third DIP, the second and third PIP, and the first carpometacarpal joints of both hands.
2. AUSCAN Function ≥ 40 aggregated points (0-100 scale)
3. Willing and able to participate in all study visits
4. Able to understand and read Danish.

Exclusion Criteria:

1. Other diseases affecting the joints of the hand (Rheumatoid arthritis, Psoriatic arthritis, ect.)
2. Widespread or generalized pain syndrome (e.g. fibromyalgia)
3. Steroid injections in the finger joints within the last month
4. Other condition that in the opinion of the investigator makes the participant unsuitable for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Change in hand physical function | Baseline, week 6 (end-of-study)
  change in physical function is measured with the Australian/Canadian Osteoarthritis Hand Index (AUSCAN).
  AUSCAN is a validated questionnaire with 3 subscales assessing pain, hand stiffness and hand function during the last 48 hours. Each question is rated on a visual analog scale from 0 (no problems) to 100 (severe problems). The subscale function will be used.

SECONDARY OUTCOMES:
Change in stiffness | Baseline, week 6
  Change in stiffness will be measured using the AUSCAN subscale stiffness, assess on a visual analogue scale (VAS) that spans from 0 (no stiffness) to 100 (worst imaginable stiffness).
Change in tender and swollen joint count | baseline, week 6
  Joint assessment includes bilateral examination of the first carpometacarpal (CMC-1), interphalangeal (IP) joint, and the second to fifth PIP (proximal interphalangeal) and DIP (distal interphalangeal) joints. The total number of swollen joints (Swollen Joint Count; SJC) and tender joints (Tender Joint Count; TJC) will be assessed for both hands by a medical doctor. The SJC and TJC will be assessed according to the European League Against Rheumatism (EULAR) handbook in a dichotomous manner.
Change in hand pain | Baseline, week 6
  A visual analogue scale (VAS) will be used to score overall hand pain. The scale spans from 0 to 100, with 0 equal no symptoms and 100 equal worst imaginable symptoms. Participants will be asked to score their average pain for the whole hand within the last week.
Change in global assessment of hand related problems | Baseline, week 6
  A visual analogue scale (VAS) will be used to score patients global assessment of hand related problems. The scale spans from 0 to 100, with 0 equal no symptoms and 100 equal worst imaginable symptoms. Participants will be asked to score their general problems related to hand function during the last week.
Change in grip strength | Baseline, week 6
  Grip strength will be assessed using the Gripp-it, an instrument that records grip force in Newtons. Three measurements will be performed on each hand and the maximum of these three measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: cecilie bartholdy, PhD, Principal Investigator — The Parker institute
Locations (1):
- Artroseambulatoriet, Frederiksberg, Denmark

REFERENCES:
- [Derived] Bartholdy C, Dossing A, Stisen ZR, Nielsen SM, Christensen R, Danneskiold-Samsoe B, Bliddal H, Henriksen M, Ellegaard K. Effect of heated mittens on physical hand function in people with hand osteoarthritis: randomised controlled trial. BMJ. 2024 Dec 17;387:e078222. doi: 10.1136/bmj-2023-078222. PMID 39689944

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04576403/SAP_000.pdf